CLINICAL TRIAL: NCT04733105
Title: Pronostic Value of Type I ANTi-Interferon Antibodies in Patients With COVID-19 Acute Respiratory Failure: a Multicenter Observational Study
Brief Title: Pronostic Value of Type I ANTi-Interferon Antibodies in Patients With COVID-19 Acute Respiratory Failure
Acronym: ANTICOV
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201254
Record Dates: First submitted 2021-01-24; First posted 2021-02-01 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-01

CONDITIONS: Acute Respiratory Failure
Keywords: COVID-19; Acute respiratory failure; ARDS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe SARS-CoV-2 infections are frequently associated with the acute respiratory distress syndrome (ARDS), which leads to a mortality of 30-40%. An altered type I interferon (IFN) response has been demonstrated in patients with severe COVID-19, together with a high viral load.

The aim of the current work is, in a large cohort of patients with severe COVID-19 admitted in the ICU, to determine the prevalence of patients with positive anti-IFN antibodies and to determine their outcome, as compared to patients having negative anti-IFN antibodies.

DETAILED DESCRIPTION:
Severe SARS-CoV-2 infections are frequently associated with the acute respiratory distress syndrome (ARDS), which leads to a mortality of 30-40%. An altered type I interferon (IFN) response has been demonstrated in patients with severe COVID-19, together with a high viral load. A recent study revealed that 10% of patients admitted in the intensive care unit (ICU) for severe COVID-19 had positive type I anti-IFN antibodies. Such finding has potentially important therapeutic implications, as patients having positive anti-IFN antibodies could benefit from targeted interventions, including plasmapheresis. The aim of the current work is, in a large cohort of patients with severe COVID-19 admitted in the ICU, to determine the prevalence of patients with positive anti-IFN antibodies and to determine their outcome, as compared to patients having negative anti-IFN antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* SARS-CoV-2 infection with a positive PCR
* Patient admitted in the ICU for acute respiratory failure (SpO2≤90% and need for supplemental oxygen or any kind of ventilator support)
* Patient or next of keen was informed of study inclusion

Exclusion Criteria:

• Patient with SARS-CoV-infection but no acute respiratory failure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with proven SARS-CoV-2 infection and acute respiratory failure admitted in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
day-28 mortality | at day-28 of intensive care unit (ICU) admission
  comparaison of day-28 mortality in patients having positive versus negative type I anti-IFN antibodies

SECONDARY OUTCOMES:
rate of positivity of type I anti-IFN antibodies | 3 months of ICU admission
  positivity of type I anti-IFN antibodies measured on a serum sample obtained at any time during ICU stay
Factors associated with type I anti-IFN antibody positivity | 24 hours of ICU admission
  Factors associated with type I anti-IFN antibody positivity available upon hospital admission, identified using uni- and multiple logistic regression analyses
hospital mortality | at day 90.
  Comparaison of hospital mortality of patients having positive versus negative type I anti-IFN antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas De PROST, MD, PhD, Study Chair — APHP
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France